CLINICAL TRIAL: NCT00002388
Title: A Study to Evaluate the Single-Dose and Steady-State Pharmacokinetics/Dynamics of 1592U89 and Its Active Moiety, 1144U88 5'-Triphosphate (1144U88-TP) Following Six Different Dosing Regimens of 1592U89 in HIV-1 Infected Subjects
Brief Title: A Study of 1592U89 in HIV-Infected Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 238G; CNAA1004
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1998-11

CONDITIONS: HIV Infections
Keywords: HIV-1; Reverse Transcriptase Inhibitors; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections | interventions — abacavir

INTERVENTIONS:
Drug: Abacavir sulfate

SUMMARY:
The purpose of this study is to see if it is safe to give 1592U89 to HIV-infected patients. This study also examines the effect 1592U89 has on plasma viral load (the level of HIV in the blood).

DETAILED DESCRIPTION:
Cohorts of 8 patients are entered sequentially into 1 of 6 1592U89 dosing regimens. All patients receive 12 weeks of monotherapy during the initial 12-week treatment phase.

On completion of the treatment phase, patients are offered continuation therapy with 1592U89 for a minimum of 12 weeks.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

Prophylaxis for opportunistic infections.

Patients must have:

* HIV-1 infection.
* CD4 cell count 100 - 500 cells/mm3 within 3 to 5 weeks prior to study drug administration.
* No active diagnosis of AIDS (other than non-visceral Kaposi's sarcoma) according to the 1993 CDC AIDS surveillance definition.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions and symptoms are excluded:

* Malabsorption syndrome or other gastrointestinal dysfunction that may interfere with drug absorption.
* Chronic disease such as diabetes, congestive heart failure, cardiomyopathy, or other cardiac dysfunction that in the opinion of the investigator, would compromise the safety of the patient.

Concurrent Medication:

Excluded:

* Immunomodulating agents.
* Chemotherapeutic agents.
* Antiretroviral therapy. NOTE:
* Patients who elect to continue study treatment into the extended phase may, after consultation with their primary physician, combine 1592U89 at a recommended dose of 300 mg bid with other licensed antiretroviral drugs.

Concurrent Treatment:

Excluded:

Radiation therapy.

Patients with the following prior conditions are excluded:

* History of clinically relevant hepatitis or pancreatitis within 6 months prior to study drug administration.
* History of hypersensitivity, anaphylactic, or idiosyncratic reaction to nucleoside analogs.

Prior Medication:

Excluded:

* Treatment with immunomodulating or cytotoxic chemotherapeutic agents within six weeks prior to study drug administration.
* Antiretroviral therapy within 2 weeks prior to administration of study drugs.

Prior Treatment:

Excluded:

Radiation therapy within six weeks prior to study drug administration. Current alcohol or illicit controlled substance use that in the opinion of the investigator, may interfere with the patient's ability to complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Evanston Hosp / Clinical Pharmacology Unit, Evanston, Illinois
  - Fenway Community Health Ctr / Research Dept, Boston, Massachusetts
  - Albany Med College / Albany Med Ctr Hosp, Albany, New York